CLINICAL TRIAL: NCT04286022
Title: Specific Neurotechnical Strength Training: Randomized Controlled Trial (NeuroTraining)
Brief Title: Specific Neurotechnical Strength Training (NeuroTraining)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, Director, Clinical Research, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NEUROTRAINING
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-02

CONDITIONS: Neuromuscular Adaptations
Keywords: Strength training; Neuromuscular adaptation
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Two randomly allocated parallel groups
Who Masked: Outcomes Assessor
Masking Description: The assessor will not be aware of the group to which each subject has been assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Speed Loss 20% Group (Experimental): The SL20% group will carry out a program based on the limitation of the speed loss, allowing to perform the exercise only until a speed loss of 20% is achieved, following a similar methodology previously published (Pareja-Blanco et al., 2017). The program will consist of a job for 4 weeks, with a frequency of 2 sessions a week. In each session, a 6-series routine with an open number of repetitions will be carried out twice, allowing as many repetitions as possible to perform until a 20% loss of execution speed is reached. The intensity of work will be 70% 1RM, resting 4 minutes between sets. As an only exercise, an elbow flexion (bicep curl) with dumbbell will be performed.
  Interventions: Other: Speed Loss 20% Strength Training
- Reduced Rest Time Group (Experimental): The RRT group will carry out a program based on the reduction of rest time between series, following a previously published methodology (Stragier et al., 2019). The program will consist of a job for 4 weeks, with a frequency of 2 sessions a week. In each session, a 5 series routine with progressive repetition volume (3 to 7) at 70% 1RM will be performed twice, resting 15 seconds between sets and 150 seconds between each of the 2 blocks. The exercise to be performed will be an elbow flexion (bicep curl) with dumbbell.
  Interventions: Other: Reduced Rest Time Strength Training

INTERVENTIONS:
Other: Speed Loss 20% Strength Training — Strength training based on the control of speed loss in execution.
  Arms: Speed Loss 20% Group
Other: Reduced Rest Time Strength Training — Strength training based on a protocol that includes reduced rest times between sets.
  Arms: Reduced Rest Time Group

SUMMARY:
This study aims to apply a novel study methodology using high density electromyography (HDEMG) to know what are the mechanisms underlying the structural and functional changes obtained by two different training methods, commonly used, facilitating their understanding, study and subsequent application according to specific needs.

DETAILED DESCRIPTION:
Different training methodologies have previously shown similar results in the improvement of structural or functional characteristics such as hypertrophy or strength. However, the different nature of their methods has suggested for years the possibility that different neuromuscular mechanisms could be behind these observed characteristics.

The development of a new technology, such as high-density electromyography (HDEMG), capable of studying new properties previously hidden from assessment methods, such as the speed of nerve impulse propagation or the frequency of motor unit discharge, has allowed a more thorough study of the mechanisms.

This study aims to apply this new study methodology to know what are the mechanisms underlying the changes at the structural and functional level obtained by two different training methods, commonly used, facilitating their understanding, study and subsequent application according to specific needs.

For this reason, the main hypothesis is the generation of different neuromuscular mechanisms and adaptations by executing, for 4 weeks, two different training methodologies, obtaining a dissociation between the results obtained at the structural level (hypertrophy), functional (generation of strength) and HDEMG analysis of the central and peripheral characteristics of the neuromuscular system in each of the programs studied.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years
* men

Exclusion Criteria:

* physical exercise that involves work of upper limbs during the time of the intervention
* upper limb injury during the previous 12 months
* systemic diseases

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Recruitment will be done only among men because of the need to use a homogeneous sample due to the heterogeneity of the test itself. Previous studies have shown a greater possibility of data analysis in men when using HDEMG.
Enrollment: 34 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Mean Discharge Rate of Brachialis Biceps Motor Units at 4 weeks | Baseline and post-intervention (4 weeks after baseline)
  The mean discharge rate of the Brachialis Biceps motor units will be evaluated using a high density electromyography device (HDEMG). For this, the signal produced during isometric contractions at different submaximal force levels (10, 30, 50, and 70%) will be recorded, using an external analog to digital signal converter Sessantaquattro (64-channel EMG amplifier; OT Bioelettronica, Turin, Italy).

SECONDARY OUTCOMES:
Speed of propagation of Brachialis Biceps Motor Units | Baseline and post-intervention (4 weeks after baseline)
  As a measure of evaluation of the peripheral characteristics of the neuromuscular system, the propagation speed of the action potentials produced by an HDEMG device will be evaluated. For this, the signal produced during isometric contractions at different submaximal force levels (10, 30, 50, and 70%) will be recorded, using the external analog to digital signal converter Sessantaquattro
Isometric force of Brachialis Biceps using hand dynamometer | Baseline and post-intervention (4 weeks after baseline)
  The isometric force at 0º, 45º and 90º will be evaluated during a maximum test of 5 seconds using a digital manual dynamometer. The peak force obtained will be obtained.
Isometric force of Brachialis Biceps using s-beam load cell | Baseline and post-intervention (4 weeks after baseline)
  The isometric force at 90º will also be evaluated through an S-type load cell (Biometrics Ltd., Newport, United Kingdom). In addition, the time needed to obtain the peak force achieved will be recorded.
Muscle thickness (thickness) of the brachial biceps using ultrasound | Baseline and post-intervention (4 weeks after baseline)
  Structural changes will be evaluated through an innocuous procedure such as ultrasound. To do this, ultrasound images will be recorded to measure the muscular and adipose thickness of the arm musculature.
Arm circumference | Baseline and post-intervention (4 weeks after baseline)
  A variable related to structural changes such as arm circumference will also be evaluated. For this, the circumference will be recorded through a measuring tape at the average distance between the acromion and the olecranon.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio I Cuesta-Vargas, PhD, Principal Investigator — University of Malaga
Locations (1):
- Health Science School , University of Malaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: Undecided